CLINICAL TRIAL: NCT05635019
Title: Food Supplementation Interventions to Improve Weight Loss for Adults With Food Insecurity and Obesity
Brief Title: FoodRx for Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 852467; R56NR020466-01 (NIH)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Food Insecurity
Keywords: obesity; food insecurity; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral weight loss counseling (BWL) alone (Active Comparator): BWL counseling alone
  Interventions: Behavioral: Behavioral weight loss counseling (BWL)
- BWL+VOUCHER (Experimental): BWL counseling and gift cards to grocery stores
  Interventions: Behavioral: BWL+VOUCHER; Behavioral: Behavioral weight loss counseling (BWL)
- BWL+HOME (Experimental): BWL counseling and home-delivered boxes of groceries
  Interventions: Behavioral: BWL+HOME; Behavioral: Behavioral weight loss counseling (BWL)

INTERVENTIONS:
Behavioral: BWL+VOUCHER — This group will receive the BWL program as well as food vouchers, in the form of grocery store gift cards. Participants will be allowed to select to receive gift cards to a grocery store or supermarket from a pre-determined list of stores. Gift cards worth $40 will be emailed or mailed to every 2 weeks after the BWL session.
  Arms: BWL+VOUCHER
Behavioral: BWL+HOME — This group will receive the BWL program as well as home-delivered boxes of groceries of low-energy density foods conducive to weight management guidelines. Groceries will include shelf-stable and perishable products like lean meats, fresh vegetables, and fruits. Every 2 weeks, participants assigned to this group will be allowed to select a choice of one of 4 boxes with slightly varied contents. Each box will have approximately $40 worth of groceries.
  Arms: BWL+HOME
Behavioral: Behavioral weight loss counseling (BWL) — The behavioral weight loss program consists of 14 individual lifestyle counseling sessions provided over 24 weeks. Each session will be approximately 15-20 minutes. Visits will be scheduled weekly for the first 4 weeks (weeks 1, 2, 3, and 4) and every-other week from weeks 6-24 (weeks 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24). The sessions will provide behavioral, dietary, and physical counseling.

SUMMARY:
This study is a 3-group, parallel design, randomized controlled trial (RCT) in 105 adults with obesity and food insecurity that will compare BWL-Alone (including standard-of-care referral and connection with community food resources; n=35) to BWL plus food supplementation with either food vouchers (BWL+VOUCHER; n=35) or home-delivered, medically tailored groceries consistent with BWL recommendations (BWL+HOME; n=35). All groups will have BWL treatment provided for 24 weeks per clinical guidelines. Food vouchers and HOME will be provided for 24 weeks of treatment. Assessments will be conducted at baseline, and weeks 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age >18 years
4. BMI >30 kg/m2 at screening visit
5. Screening positive for food insecurity using a score of >3 on the 10-item US Adult Food Security Survey Module109
6. Completion of baseline assessments
7. Ability to engage in physical activity (i.e., can walk at least 2 blocks)
8. Willing and able to provide pictures of food receipts to study team (or mail actual receipts)
9. Ability to reliably receive packages at a consistent location in a timely manner
10. Telephone or internet service to communicate with study staff
11. For females of reproductive potential: agreement to use of highly effective contraception for during study participation

Exclusion Criteria:

1. Serious medical conditions (e.g., type 1 or type 2 diabetes, renal failure) that may pose a risk to the participant during intervention, cause a change in weight, or limit ability to adhere to the program's behavioral recommendations
2. Significant psychiatric conditions (e.g., active substance abuse, schizophrenia) that may pose a risk to the participant during intervention, cause a change in weight, or limit ability to adhere to the program's behavioral recommendations
3. Breastfeeding, pregnant or planning pregnancy in the next 6 months
4. Planned move from the Philadelphia area in the next 6 months
5. Weight loss of >5 kg in the previous 90 days
6. Recently began a course of or changed the dosage of medication that can cause significant weight change (±5 kg)
7. Previous or planned obesity treatment with surgery (excluding lap band if removed for >1 year) or a weight-loss device
8. Use of prescription or over the counter medications for chronic weight management in the past 3 months
9. Household member already participating in study due to potential contamination effects
10. Lack of stable residence and ability to store and prepare food

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phone screen. Interested participants were consented verbally over the phone by study staff to participate in the initial telephone screening.
  Eligible participants attended a 1.5-hour, in-person screening visit.
Period: Overall Study
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+VOUCHER | BWL+HOME
Started | 35 | 35 | 35
Completed | 35 | 35 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+VOUCHER | BWL+HOME | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-reported age at enrollment
  years | 49.7 (14.8) | 55.4 (11.3) | 53.3 (15.0) | 52.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 31 | 92
  Male | 5 | 4 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 27 | 26 | 76
  White | 8 | 7 | 8 | 23
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Baseline weight (kg) [Mean (Standard Deviation); unit: kg] — Baseline body weight (kg)
  kg | 108.0 (17.9) | 104.6 (24.8) | 110.4 (17.1) | 107.7 (20.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Body Weight at 24 Weeks (BWL+VOUCHER and BWL+HOME vs BWL-Alone)
Description: Comparison of BWL+VOUCHER and BWL+HOME vs BWL-Alone in weight change (percent of initial weight) at 24 weeks. Positive numbers represent increases and negative numbers represent decreases.
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: Percent initial weight loss
Groups:
- BWL+Supplement (BWL+VOUCHER or BWL+HOME): BWL counseling and gift cards to grocery stores or BWL counseling and home-delivered boxes of groceries
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+Supplement (BWL+VOUCHER or BWL+HOME)
Number analyzed (Participants) | 35 | 70
Percent initial weight loss | -2.7 (0.5) | -3.0 (0.3)

2. Secondary Outcome: Percent Change in Total Body Weight at 24 Weeks (BWL+HOME vs BWL+VOUCHER)
Description: Comparison of BWL+HOME vs BWL+VOUCHER in weight loss (percent of initial weight) at 24 weeks. Negative values indicate losses. Positive values indicate gains.
Time Frame: Change from baseline to 24 weeks
Measure: Mean (Standard Error); unit: Percent initial weight loss
Arm/Group | BWL+VOUCHER | BWL+HOME
Number analyzed (Participants) | 35 | 35
Percent initial weight loss | -3.5 (0.4) | -2.7 (0.5)

3. Secondary Outcome: General Health-related Quality of Life (BWL+VOUCHER and BWL+HOME vs BWL-Alone)
Description: Change from baseline to week 24 in general health-related quality of life (physical function component score) as assessed with the Short Form-36. Scores range from 0 (worse) to 100 (best).
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+Supplement (BWL+VOUCHER or BWL+HOME)
Number analyzed (Participants) | 35 | 35
score on a scale | -0.5 (2.0) | -0.64 (1.3)

4. Secondary Outcome: Weight-related Quality of Life (BWL+VOUCHER and BWL+HOME vs BWL-Alone)
Description: Change from baseline to week 24 in weight-related quality of life as assessed with the Impact of Weight on Quality of Life-Lite. Scores range from 0 (worse) to 100 (best).
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+Supplement (BWL+VOUCHER or BWL+HOME)
Number analyzed (Participants) | 35 | 35
score on a scale | 7.8 (2.5) | 8.8 (1.6)

5. Secondary Outcome: Dietary Quality as Assessed by Skin Carotenoid Levels (BWL+VOUCHER and BWL+HOME vs BWL-Alone)
Description: Change from baseline to week 24 in skin carotenoid levels (skin carotenoids are measured on a scale from 0-800). Lower scores are worse and higher scores indicate a better outcome.
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+Supplement (BWL+VOUCHER or BWL+HOME)
Number analyzed (Participants) | 35 | 35
units on a scale | 15.6 (10.3) | 7.1 (6.7)

6. Secondary Outcome: Dietary Quality as Assessed by the Healthy Eating Index (BWL+VOUCHER and BWL+HOME vs BWL-Alone)
Description: Change from baseline to week 24 in Healthy Eating Index scores as measured with the Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool. Scores range from 0 (worse) to 100 (best).
Time Frame: Change from baseline to 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+VOUCHER | BWL+HOME
Number analyzed (Participants) | 35 | 35 | 35
score on a scale | 0.4 (3.0) | 10.8 (2.8) | .8 (2.8)

7. Secondary Outcome: General Health-related Quality of Life (BWL+VOUCHER vs BWL+HOME)
Description: Change from baseline to week 24 in general health-related quality of life as assessed with the Short Form-36. Scores range from 0 (worse) to 100 (best).
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BWL+VOUCHER | BWL+HOME
Number analyzed (Participants) | 35 | 35
score on a scale | 0.4 (1.8) | -1.6 (1.8)

8. Secondary Outcome: Weight-related Quality of Life (BWL+VOUCHER vs BWL+HOME)
Description: Change from baseline to week 24 in weight-related quality of life (physical component scale) as assessed with the Impact of Weight on Quality of Life-Lite. Scores range from 0 (worse) to 100 (best).
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BWL+VOUCHER | BWL+HOME
Number analyzed (Participants) | 35 | 35
score on a scale | 0.4 (1.8) | -1.6 (1.8)

9. Secondary Outcome: Dietary Quality as Assessed by Skin Carotenoid Levels (BWL+VOUCHER vs BWL+HOME)
Description: as for outcome 5
Time Frame: Change from baseline to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BWL+VOUCHER | BWL+HOME
Number analyzed (Participants) | 35 | 35
units on a scale | 16.2 (8.6) | -1.6 (8.5)

10. Secondary Outcome: Dietary Quality as Assessed by the Healthy Eating Index (BWL+VOUCHER vs BWL+HOME)
Description: Change from baseline to week 24 in Healthy Eating Index scores as measured with the ASA24. Scores range from 0 (worse) to 100 (best).
Time Frame: Change from baseline to 24 weeks
Population: Intention to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BWL+VOUCHER | BWL+HOME
Number analyzed (Participants) | 35 | 35
score on a scale | 10.8 (2.8) | .8 (2.8)

ADVERSE EVENTS:
Time Frame: Baseline to 24 weeks
Description: As per clinicaltrials.gov
Arm/Group | Behavioral Weight Loss Counseling (BWL) Alone | BWL+VOUCHER | BWL+HOME
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT05635019/Prot_SAP_000.pdf